CLINICAL TRIAL: NCT02387294
Title: Immunogenicity and Tolerability Study of Fluval AB Novo Suspension for Injection (Trivalent, Seasonal Influenza Vaccine, Active Ingredient Content: 6 μg HA/Strain/0.5 ml) for Children and Adolescents
Brief Title: Immunogenicity and Tolerability Study of Fluval AB Novo Suspension for Injection for Children and Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fluart Innovative Vaccine Ltd, Hungary (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FABNovo-H-16
Record Dates: First submitted 2014-10-16; First posted 2015-03-13 (Estimated); Results first posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2015-03

CONDITIONS: Human Influenza
Keywords: immunogenicity; reduced dose; Phase III; tolerability; safety
MeSH Terms: conditions — Influenza, Human | interventions — Vaccination; Injections

STUDY DESIGN:
Intervention Model Description: parallel-group study in two paediatric age groups
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Age group 1: children (3-11 years) (Experimental): Intervention: Vaccination with Fluval AB Novo suspension for injection.
  Dosage: Half dose of a single dose (0.25 ml) vaccine, administered intramuscularly.
  Interventions: Biological: Vaccination with Fluval AB Novo suspension for injection, half dose of a single intramuscular dose (0.25 ml)
- Age group 2: adolescents (12-18 years) (Experimental): Intervention: Vaccination with Fluval AB Novo suspension for injection.
  Dosage: A single dose (0.5 ml) vaccine, administered intramuscularly.
  Interventions: Biological: Vaccination with Fluval AB Novo suspension for injection, single intramuscular dose (0.5 ml)

INTERVENTIONS:
Biological: Vaccination with Fluval AB Novo suspension for injection, half dose of a single intramuscular dose (0.25 ml) — vaccination
  Other Names: Fluval AB Novo suspension for injection
  Arms: Age group 1: children (3-11 years)
Biological: Vaccination with Fluval AB Novo suspension for injection, single intramuscular dose (0.5 ml) — vaccination
  Arms: Age group 2: adolescents (12-18 years)

SUMMARY:
Immunogenicity and Tolerability Study of Fluval AB Novo Suspension for Injection (trivalent, seasonal influenza vaccine, active ingredient content: 6 μg HA/strain/0.5 ml) for Children and Adolescents.

DETAILED DESCRIPTION:
STUDY PERIOD:

Length of enrollment: 2 weeks (estimated) Participation per subject: max. 1 month

OBJECTIVES:

Immunogenicity Objectives:

To assess immunogenicity of a single intramuscular injection of Fluval AB Novo suspension for injection (trivalent, seasonal influenza vaccine, active ingredient content: 6 μg HA/0.5 ml of seasonal A/H1N1, A/H3N2 and B influenza antigens each), as measured by haemagglutination inhibition (HI) test.

Safety and Tolerability Objectives:

To evaluate safety and tolerability (incidence of adverse events) of a single intramuscular injection of Fluval AB Novo suspension for injection.

CLINICAL PHASE:

Phase III

TYPE:

Interventional, prevention

DESIGN:

Non-controlled, open, multi-centre

METHODS:

In this uncontrolled, open, multi-centre immunogenicity and tolerability study subjects were enrolled into two groups according to age:

Age group 1: children (3-11 years): single intramuscular injection of Fluval AB Novo 0.25 ml suspension for injection; Age group 2: adolescents (12-18 years): single intramuscular injection of Fluval AB Novo 0.5 ml suspension for injection; Subjects were observed for 30 minutes after the injection for any immediate reactions.

All adolescent subjects aged 12 to 18 years and the legitimate representatives of all volunteers were requested to complete a Diary Card (DC) to record local reactions (injection site pain, erythema, swelling, induration, numbness, sensitivity and haematoma) and systemic reactions (fever, shivering, headache, malaise, fatigue, sweating, nausea, myalgia, arthralgia, dizziness and urticaria) starting on the day of vaccination on Visit 1 (Day 0) until 7 days following that.

All adverse events were collected during the period of Visit 1 (Day 0) to Visit 2 (between Day 21 and Day 28); Serum samples for immunogenicity assays were collected immediately before immunization on Visit 1 (Day 0) and on Visit 2 (between Day 21 and Day 28) in all subjects. Immunogenicity were evaluated by HI test.

INVESTIGATIONAL MEDICINAL PRODUCT:

Fluval AB Novo suspension for injection (trivalent, seasonal influenza vaccine, active ingredient content: 6 μg HA/0.5 ml of seasonal A/H1N1, A/H3N2 and B influenza antigens each) with aluminium phosphate gel adjuvant.

Lot No.: FL-N-05/13

CONCOMITANT VACCINES:

No concomitant vaccination is permitted for the duration of the study except for post-exposure vaccination in a medical emergency (e.g. tetanus, rabies, hepatitis).

STUDY POPULATION:

Considering approximately 17% of drop-out (one participant out of six), in total 120 subjects (60 subjects in each age group) were enrolled in order to achieve at least 100 evaluable subjects (50 subjects in each age group).

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 to 11 years, adolescents aged 12 to 18 years from both sexes;
* Are in good health (as determined by vital signs and existing medical condition) or are in stable medical condition. Subjects will not be excluded with known adequately treated clinically significant organ or systemic diseases (e.g. asthma or diabetes), such that, in the opinion of the investigator, the significance of the disease will not compromise the subject's participation in the study;
* Female volunteers of childbearing potential with a negative result from the urine pregnancy test prior to vaccination who agrees to use an acceptable contraception method or abstinence throughout the trial and not become pregnant for the duration of the study;
* Capability of adolescent participants aged 12 to 18 years and the legitimate representative of all volunteers to understand and comply with planned study procedures;
* Adolescent participants aged 12 to 18 years and the legitimate representative of all volunteers provide written Informed Consent (IC) prior to initiation of study procedures;
* Absence of existence of any exclusion criteria.

Exclusion Criteria:

* Pregnancy, breast feeding or positive urine pregnancy test at baseline prior to vaccination. Female subjects who are able to bear children but not willing to use an acceptable contraception method for the duration of the study.
* Known hypersensitivity to eggs, thiomersal, formaldehyde, gentamycin, ciprofloxacin, neomycin, vancomycin or any other component of the vaccine;
* History of Guillain-Barré syndrome;
* History of neurological symptoms or signs, or anaphylactic shock following administration of any vaccine;
* Serious disease, such as cancer, autoimmune disease, advanced arteriosclerotic disease, complicated diabetes mellitus, acute or progressive hepatic disease, acute or progressive renal disease, congestive heart failure;
* Immunosuppressive therapy within 36 months prior to vaccination;
* Concomitant corticosteroid therapy, including high-dose inhaled corticosteroids;
* Receipt of immunostimulants,
* Receipt of parenteral immunoglobulin, blood products and/or plasma derivate within 3 months prior to vaccination;
* Suspected or known HIV, HBV or HCV infection;
* Acute disease and/or axillary temperature ≥37oC within 3 days prior to vaccination;
* Vaccine therapy within 4 weeks prior to vaccination;
* Influenza vaccination (any kind) within 6 months prior to vaccination;
* Experimental drug therapy within 4 weeks prior to vaccination;
* Concomitant participation in another clinical study;
* Any condition which, in the opinion of the investigator, may interfere with the evaluation of the study;
* Past or current psychiatric disease of the volunteer or the legitimate representative that upon judgement of the investigator may have effect on the objective decision-making of the volunteer;
* Alcohol or drug abuse of the participant or the legitimate representative.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Age Group 1: Children (3-11 Years): Intervention: Vaccination with Fluval AB Novo
  Dosage: half of the single dose
- Age Group 2: Adolescents: Intervention: Vaccination with Fluval AB Novo
  Dosage: single dose
Period: Overall Study
Arm/Group | Age Group 1: Children (3-11 Years) | Age Group 2: Adolescents
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Age Group 1: Children (3-11 Years) | Age Group 2: Adolescents (12-18 Years) | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 60 | 60 | 120
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Standard Deviation); unit: years] — Age at the time of enrolment
  years | 7.93 (2.65) | 14.38 (1.54) | 11.16 (3.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 30 | 53
  Male | 37 | 30 | 67
Region of Enrollment [Count of Participants; unit: Participants]
  Hungary | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Increase in Geometric Mean Titre Ratio, A/H1N1 Strain
Description: Ratio of Day 0 and Day 21-28 antihaemagglutination inhibition titres
  Requirement: > 2.5
Time Frame: 21-28 days after vaccination
Population: PP population (subjects whose antihaemagglutination inhibition titres are available both Day 0 and Day 21-28 visits)
Measure: Mean (95% Confidence Interval); unit: Ratio of Day 0 and Day 21-28 titres
Groups:
- Age Group 2: Adolescents: Intervention: Vaccination with Fluval AB Novo suspension for injection.
  Dosage: A single dose (0.5 ml) vaccine, administered intramuscularly.
Arm/Group | Age Group 1: Children (3-11 Years) | Age Group 2: Adolescents
Number analyzed (Participants) | 60 | 60
Ratio of Day 0 and Day 21-28 titres | 4.337 [3.432 to 5.480] | 4.702 [3.595 to 6.151]

2. Primary Outcome: Increase in Geometric Mean Titre Ratio, A/H3N2 Strain
Description: Ratio of Day 0 and Day 21-28 antihaemagglutination inhibition titres
  Requirement: > 2.5
Time Frame: 21-28 days after vaccination
Population: PP population (subjects whose antihaemagglutination inhibition titres are available both Day 0 and Day 21-28 visits)
Measure: Mean (95% Confidence Interval); unit: Ratio of Day 0 and Day 21-28 antihaemagg
Arm/Group | Age Group 1: Children (3-11 Years) | Age Group 2: Adolescents (12-18 Years)
Number analyzed (Participants) | 60 | 60
Ratio of Day 0 and Day 21-28 antihaemagg | 4.982 [3.847 to 6.451] | 5.993 [4.207 to 8.539]

3. Primary Outcome: Increase in Geometric Mean Titre Ratio, B Strain
Description: Ratio of Day 0 and Day 21-28 antihaemagglutination inhibition titres
  Requirement: > 2.5
Time Frame: 21-28 days after vaccination
Population: PP population (subjects whose antihaemagglutination inhibition titres are available both Day 0 and Day 21-28 visits)
Measure: Mean (95% Confidence Interval); unit: Ratio of Day 0 and Day 21-28 titres
Arm/Group | Age Group 1: Children (3-11 Years) | Age Group 2: Adolescents (12-18 Years)
Number analyzed (Participants) | 60 | 60
Ratio of Day 0 and Day 21-28 titres | 4.262 [3.383 to 5.370] | 4.757 [3.762 to 6.014]

4. Primary Outcome: Seroconversion, A/H1N1 Strain
Description: Proportion of subjects seroconverted or had a significant increase in titres
  Requirement: > 40 %
Time Frame: 21-28 days after vaccination
Population: PP population (subjects whose antihaemagglutination inhibition titres are available both Day 0 and Day 21-28 visits)
Measure: Number; unit: percentage of subjects seroconverted
Arm/Group | Age Group 1: Children (3-11 Years) | Age Group 2: Adolescents (12-18 Years)
Number analyzed (Participants) | 60 | 60
percentage of subjects seroconverted | 61.67 | 66.67

5. Primary Outcome: Seroconversion, A/H3N2 Strain
Description: Proportion of subjects seroconverted or had a significant increase in titres
  Requirement: > 40 %
Time Frame: 21-28 days after vaccination
Population: PP population (subjects whose antihaemagglutination inhibition titres are available both Day 0 and Day 21-28 visits)
Measure: Number; unit: percentage of subjects seroconverted
Arm/Group | Age Group 1: Children (3-11 Years) | Age Group 2: Adolescents (12-18 Years)
Number analyzed (Participants) | 60 | 60
percentage of subjects seroconverted | 58.33 | 61.67

6. Primary Outcome: Seroconversion, B Strain
Description: Proportion of subjects seroconverted or had a significant increase in titres
  Requirement: > 40 %
Time Frame: 21-28 days after vaccination
Population: PP population (subjects whose antihaemagglutination inhibition titres are available both Day 0 and Day 21-28 visits)
Measure: Number; unit: percentage of subjects seroconverted
Arm/Group | Age Group 1: Children (3-11 Years) | Age Group 2: Adolescents (12-18 Years)
Number analyzed (Participants) | 60 | 60
percentage of subjects seroconverted | 66.67 | 70.00

7. Primary Outcome: Seroprotection, A/H1N1 Strain
Description: Proportion of subjects seroprotected
  Requirement: > 70 %
Time Frame: 21-28 days after vaccination
Population: PP population (subjects whose antihaemagglutination inhibition titres are available both Day 0 and Day 21-28 visits)
Measure: Number; unit: percentage of subjects seroprotected
Arm/Group | Age Group 1: Children (3-11 Years) | Age Group 2: Adolescents (12-18 Years)
Number analyzed (Participants) | 60 | 60
percentage of subjects seroprotected | 91.67 | 96.67

8. Primary Outcome: Seroprotection, A/H3N2 Strain
Description: Proportion of subjects seroprotected
  Requirement: > 70 %
Time Frame: 21-28 days after vaccination
Population: PP population (subjects whose antihaemagglutination inhibition titres are available both Day 0 and Day 21-28 visits)
Measure: Number; unit: percentage of subjects seroprotected
Arm/Group | Age Group 1: Children (3-11 Years) | Age Group 2: Adolescents (12-18 Years)
Number analyzed (Participants) | 60 | 60
percentage of subjects seroprotected | 95.00 | 95.00

9. Primary Outcome: Seroprotection, B Strain
Description: Proportion of subjects seroprotected
  Requirement: > 70 %
Time Frame: 21-28 days after vaccination
Population: PP population (subjects whose antihaemagglutination inhibition titres are available both Day 0 and Day 21-28 visits)
Measure: Number; unit: percentage of subjects seroprotected
Arm/Group | Age Group 1: Children (3-11 Years) | Age Group 2: Adolescents (12-18 Years)
Number analyzed (Participants) | 60 | 60
percentage of subjects seroprotected | 80.00 | 86.67

ADVERSE EVENTS:
Time Frame: 21-28 days after vaccination
Description: Diary card was used by all subjects to record Adverse Events between Day 0-7 (during 7 days after vaccination), afterwards, Adverse Events were recorded on Day 21-28. Serious Adverse Events were reported in 24 hours after its occurrence.
Arm/Group | Age Group 1: Children (3-11 Years) | Age Group 2: Adolescents (12-18 Years)
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 59/60 | 56/60
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Age Group 1: Children (3-11 Years) (N=60) | Age Group 2: Adolescents (12-18 Years) (N=60)
vaccination site pain (General disorders) | 21 (21) | 17 (17) — pain at the vaccination site
vaccination site erythema (General disorders) | 7 (7) | 2 (2) — erythema at the vaccination site
vaccination site swelling (General disorders) | 7 (7) | 2 (2) — swelling at the vaccination site
myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 8 (8) — myalgia
malaise (General disorders) | 2 (2) | 7 (7) — malaise
vaccination site induration (General disorders) | 3 (3) | 5 (5) — induration at vaccination site
vaccination site haematoma (General disorders) | 2 (2) | 0 (0) — haematoma at vaccination site
chills (General disorders) | 2 (2) | 1 (1) — chills
pharyngitis (Infections and infestations) | 1 (1) | 0 (0) — pharyngitis
helminthic infection (Infections and infestations) | 1 (1) | 0 (0) — helminthic infection
headache (Nervous system disorders) | 0 (0) | 5 (5) — headcahe
hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) — allergic reaction
cystitis (Infections and infestations) | 0 (0) | 1 (1) — cystitis
pyrexia (General disorders) | 3 (3) | 3 (3) — fever
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — cough
vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) — vomiting
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — abdominal pain
syncope (Nervous system disorders) | 2 (2) | 1 (1) — collapsus
nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) — common cold
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) — sore throat

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that the sponsor in the frames of the general confidentiality agreement is that the PI cannot release any information concenning the study without the prior consent of the sponsor. To further specification is provided.